CLINICAL TRIAL: NCT06889051
Title: Comparison Study Between Using Retrograde Flexible Ureteroscopy With Flexible & Navigable Suction Ureteral Access Sheath Versus Retrograde Flexible Ureteroscopy With Antegrade Suction in Lower Calyceal Stone: A Randomized Controlled Trial
Brief Title: Comparison of Flexible & Navigable Suction Ureteral Access Sheath vs. Antegrade Suction in Retrograde Flexible Ureteroscopy for Lower Calyceal Stones
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tamer Abd El-Wahab Diab, Lecturer of Urology, Faculty of Medicine., Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-290-2025
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Nephrolithiasis; Urolithiasis; Endourology
Keywords: Flexible Ureteroscopy (FURS); Ureteral Access Sheath (UAS); Suction Ureteral Access Sheath (FANS); Antegrade Suction; Percutaneous Nephrostomy (PCN); Laser Lithotripsy
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial comparing two different suction techniques during retrograde flexible ureteroscopy (FURS) for lower calyceal renal stones. Participants will be assigned to one of two groups:
  * Group A (Intervention Group) - flexible ureteroscopy (FURS) with Flexible & Navigable Suction Ureteral Access Sheath (FANS)
  * Group B (Control Group) - flexible ureteroscopy (FURS) with Antegrade Suction via percutaneous nephrostomy.
  The study will assess stone-free rates (SFR), operative time, and complications.
Masking Description: This is an open-label trial with no masking, as both the surgeon and patient will be aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible & Navigable Suction Ureteral Access Sheath (FANS) Group (Experimental): Patients in this group will undergo retrograde flexible ureteroscopy (FURS) with the Flexible & Navigable Suction Ureteral Access Sheath (FANS). The FANS facilitates continuous suctioning, improving stone fragment evacuation, reducing intrarenal pressure, and optimizing stone-free rates (SFR).
  Interventions: Procedure: Flexible & Navigable Suction Ureteral Access Sheath (FANS)
- Antegrade Suction with Flexible Ureteroscopy (FURS) Group (Active Comparator): Patients in this group will undergo retrograde flexible ureteroscopy (FURS) with antegrade suction, using a percutaneous nephrostomy (PCN) access for suctioning from the kidney during the procedure. This method aims to enhance stone fragment clearance and reduce intrarenal pressure without using a ureteral access sheath.
  Interventions: Procedure: Antegrade Suction via Percutaneous Nephrostomy

INTERVENTIONS:
Procedure: Flexible & Navigable Suction Ureteral Access Sheath (FANS) — The Flexible & Navigable Suction Ureteral Access Sheath (FANS) is used during retrograde flexible ureteroscopy (FURS) for renal stones (1.5-2 cm). It allows continuous active suctioning, improving stone fragment evacuation, reducing operative time, lowering intrarenal pressure, and optimizing stone-free rates (SFR). The procedure involves inserting the Navigator 10F, 55 cm YIGAOMED FANS over a guidewire, followed by flexible ureteroscopy with PUSEN® 9.2 Fr ureteroscope and laser lithotripsy using Holmium Laser (JenaSurgical® MultiPulse HoPLUS™ 150W).
  Arms: Flexible & Navigable Suction Ureteral Access Sheath (FANS) Group
Procedure: Antegrade Suction via Percutaneous Nephrostomy — This technique involves antegrade suction from the kidney during flexible ureteroscopy (FURS) without the use of a ureteral access sheath. A percutaneous nephrostomy (PCN) tract is created using an 18G needle, and a 6F renal dilator is placed and fixed to the skin, allowing for direct suctioning from the collecting system. Following this, retrograde flexible ureteroscopy (FURS) is performed using the PUSEN® 9.2 Fr ureteroscope and Holmium Laser (JenaSurgical® MultiPulse HoPLUS™ 150W) for stone fragmentation. This technique aims to improve stone clearance while minimizing ureteral trauma associated with access sheaths.
  Arms: Antegrade Suction with Flexible Ureteroscopy (FURS) Group

SUMMARY:
This randomized controlled trial aims to compare the efficacy and safety of two suction techniques during retrograde flexible ureteroscopy (FURS) for lower calyceal renal stones measuring 1.5-2 cm. The study evaluates Flexible & Navigable Suction Ureteral Access Sheath (FANS) versus Antegrade Suction (via percutaneous access) in improving stone-free rates (SFR), reducing operative time, and minimizing complications such as bleeding, ureteral injury, and infection. A total of 120 adult patients will be randomized into two groups, undergoing either flexible ureteroscopy (FURS) with Flexible & Navigable Suction Ureteral Access Sheath (FANS) or flexible ureteroscopy (FURS) with antegrade suction, at Banha University Faculty of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Patients diagnosed with renal stones (1.5-2 cm) confirmed by non-contrast computed tomography (NCCT)
* Patients undergoing flexible ureteroscopy (FURS) as the primary treatment approach
* Patients with no active urinary tract infection (UTI) at baseline
* Patients who provide written informed consent

Exclusion Criteria:

* Patients with anatomical anomalies (e.g., horseshoe kidney, PUJ obstruction)
* Patients with a single functioning kidney
* Pregnant women
* Patients with a history of urological malignancy
* Patients with active bleeding disorders or those on anticoagulant therapy that cannot be safely discontinued
* Patients at high risk for anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Stone-Free Rate (SFR) | 1 Month Postoperative
  The stone-free rate (SFR) will be assessed one month postoperatively using non-contrast computed tomography (NCCT) to determine the presence or absence of residual stone fragments ≥4 mm. A higher SFR indicates better effectiveness of the intervention.

SECONDARY OUTCOMES:
Operative Time | During Surgery
  The total operative time will be recorded from the initial endoscopic access to procedure completion. This includes access sheath insertion, ureteroscopy, lithotripsy, and final stone evacuation. A shorter operative time is indicative of a more efficient technique.
Intraoperative Bleeding Requiring Intervention | During Surgery
  The incidence of ureteral injuries, including mucosal damage, perforation, or full-thickness injury, will be documented. The severity will be graded based on endoscopic findings and clinical impact.
Ureteral Injury | During Surgery
  The incidence of ureteral injuries, including mucosal damage, perforation, or full-thickness injury, will be documented. The severity will be graded based on endoscopic findings and clinical impact.
Postoperative Hematuria | Within 7 Days Postoperative
  The presence of postoperative hematuria (macroscopic bleeding) will be assessed. It will be classified as mild (self-limited), moderate (requiring irrigation), or severe (requiring intervention such as transfusion or embolization).
Postoperative Urosepsis | Within 7 Days Postoperative
  The incidence of postoperative urosepsis, defined as systemic inflammatory response syndrome (SIRS) with a positive urine culture and clinical deterioration requiring IV antibiotics or ICU admission, will be recorded.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including baseline characteristics, intraoperative details, postoperative outcomes, and complication data for research purposes. No personally identifiable information will be disclosed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: * Start Date: Upon publication of primary study results
  * End Date: Available for 5 years after study completion